CLINICAL TRIAL: NCT01209182
Title: In Vitro Detection of Tissue Abnormality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LS BioPath (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSB-01
Record Dates: First submitted 2010-09-21; First posted 2010-09-27 (Estimated); Last update posted 2022-10-03 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Intervention Model Description: 2 phase study: Phase 1 - Validation of safety and accuracy when used ex-vivo to image excised breast surgery specimens Phase 2 - To guide surgeon's decision to re-excise additional margins during primary operation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Device image reading (Experimental): Tissue images generated by the device are read by surgeons to determine if the tissue area under test has abnormal component or not. When Images generated by the device are read by surgeons as abnormal an additional margin of tissue is removed. The new margin is also imaged by the device to ensure complete tumor excision.
  Interventions: Device: Testing a new device (LS BioPath TOUCH) on excised tissue

INTERVENTIONS:
Device: Testing a new device (LS BioPath TOUCH) on excised tissue — Measurements are obtained with test device on excised tissue.

SUMMARY:
Intraoperative ex-vivo use of the ClearEdge Imaging Device in Breast Conserving Surgery to image the excised tissue surgical margins. The study is designed to demonstrate reduction in the need for repeat surgeries after breast conserving surgeries by using the ClearEdge as an adjunct imaging device to the standard of care.

DETAILED DESCRIPTION:
Intraoperative real-time margin assessment of breast conserving surgeries can reduce the need for repeat operations due to cancer involved margins. Repeat operations result in excessive removal of benign tissue, increased risk for infection, slower healing and inferior cosmetic results. In the current standard of care, the status of the margins is determined by pathology only several days after surgery. An intraoperative assessment of the margins enables complete tumor excision in a single surgery.

The proposed randomized controlled study will evaluate the benefits of adding the ClearEdge imaging device to the Standard of Care (SoC) of margins assessment in breast conserving surgeries. The study will assess whether there is an improvement in the detection of cancer involved margins by measuring whether removal at the time of primary surgical treatment can reduce the need for repeat surgeries as compared to the SoC, which does not use the device.

ClearEdge is a CE marked device already been used in several hospitals in the UK. It was used in a prospective single arm and 2 phases clinical study. It was demonstrated that surgeons successfully used the device to identify cancer involved margins and that it can reduce the need for repeat surgeries by meeting the margins depth criteria to require repeat operations. European Journal of Oncology Surgery. 2016; 42 (12): 1834-1840. In addition, the device was clinically evaluated by several hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 25-80 who are scheduled for surgical excision of tissue.

Exclusion Criteria:

* No prior history of surgery at location of current surgery.

Ages: 25 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — biologic females
Enrollment: 121 (Actual)
Dates: Start 2010-10-15 (Actual); Primary Completion 2011-12-13 (Actual); Study Completion 2012-01-09 (Actual)

PRIMARY OUTCOMES:
•Accuracy of LS BioPath TOUCH device compared to pathology | 1 week after surgery
  Assess percentage of FP and FN of test device results compared to pathology results

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lagios, MD, Principal Investigator — St. Mary's Medical Center
Locations (1):
- St. Mary's, San Francisco, California, United States